CLINICAL TRIAL: NCT05508737
Title: Open-label Phase II Study With Lead-in Safety Cohort of Pembrolizumab (Keytruda®) and Trifluridine/Tipiracil (Lonsurf®) Combination Treatment in Patients With Previously Treated Advanced Gastric Cancer
Brief Title: Pembrolizumab and Trifluridine/Tipiracil With Previously Treated Advanced Gastric Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, Severance Hospital, Yonsei University Health System, Yonsei University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0582
Record Dates: First submitted 2022-07-07; First posted 2022-08-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gastric and Gastroesophageal Junction Adenocarcinoma
Keywords: Pembrolizumab(Keytruda®); Trifluridine/Tipiracil (Lonsurf®)
MeSH Terms: interventions — pembrolizumab; Trifluridine; tipiracil; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IO experienced (Experimental): Pembrolizumab 400 mg every 6 weeks (Q6W), trifluridine/tipiracil at 35 or 30 mg/m2 twice daily (BID) for 5 days a week (D1-5, D8-12) with 2 days rest for 2 weeks, followed by a 14-day rest, repeated every 4 weeks (Q4W)
  Interventions: Drug: Pembrolizumab (Keytruda®), Trifluridine/Tipiracil (Lonsurf®)
- IO non-experienced (Experimental): Pembrolizumab 400 mg every 6 weeks (Q6W), trifluridine/tipiracil at 35 or 30 mg/m2 twice daily (BID) for 5 days a week (D1-5, D8-12) with 2 days rest for 2 weeks, followed by a 14-day rest, repeated every 4 weeks (Q4W)
  Interventions: Drug: Pembrolizumab (Keytruda®), Trifluridine/Tipiracil (Lonsurf®)

INTERVENTIONS:
Drug: Pembrolizumab (Keytruda®), Trifluridine/Tipiracil (Lonsurf®) — arms : Pembrolizumab 400 mg every 6 weeks (Q6W), trifluridine/tipiracil at 35 or 30 mg/m2 twice daily (BID) for 5 days a week (D1-5, D8-12) with 2 days rest for 2 weeks, followed by a 14-day rest, repeated every 4 weeks (Q4W)
  Other Names: Pembrolizumab (Keytruda®); Trifluridine/Tipiracil (Lonsurf®)

SUMMARY:
This is a two-part, Phase II, open-label, single arm, multi-center study to determine the efficacy of pembrolizumab in combination with TAS-102 (trifluridine/tipiracil) in patients with advanced gastric cancer who have progressed after prior treatment with or without anti-PD-1/PD-L1 agent, and to further assess the safety and tolerability of this combination treatment.

DETAILED DESCRIPTION:
This is a two-part, Phase II, open-label, single arm, multi-center study to determine the efficacy of pembrolizumab in combination with TAS-102 (trifluridine/tipiracil) in patients with advanced gastric cancer who have progressed after prior treatment with or without anti-PD-1/PD-L1 agent, and to further assess the safety and tolerability of this combination treatment. In lead-in-safety cohort, recommended dose of trifluridine/tipiracil combined with pembrolizumab will be determined with dose-limiting toxicity (DLT) and safety. Pembrolizumab dose will be fixed with current recommended dose of 400mg IV every 6 weeks (Q6W). There will be 2 dose cohort for trifluridine/tipiracil; dose level 1 is trifluridine/tipiracil 35mg/m2 BID, D1-5, D8-12, every 4 weeks (Q4W) and dose level 0 is trifluridine/tipiracil 30mg/m2 BID, D1-5, D8-12, every 4 weeks (Q4W). DLT will be evaluated during first 6 weeks. In the subsequent expansion Phase II part, patients will be recruited from four sites to evaluate the efficacy and safety of the combination therapy in 2 cohorts, anti-PD-1/PD-L1 inhibitor naive and exposure cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent fo the trial.
2. Is male or female at least 18 years of age.
3. Has a histologically or cytologically confirmed diagnosis of advanced or metastatic gastric/gastroesophageal junction (GEJ) adenocarcinoma.
4. Has previously received at least 2 prior regiments.
5. Has a life expectancy of at least 3 months.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Have 1 or more measurable disease as determined by RECIST 1.1.
8. Is able to take medications orally.
9. Has adequate organ function as defined by the following criteria.
10. Is willing to follow and follow research procedures.
11. A male participant must agree to use a contraception of this protocol during the treatment period and for at least 120 days post TAS-102.
12. A female participant is eligible to participate if she is not pregnant or breastfeeding.

Exclusion Criteria:

1. Has other concurrently active malignancies.
2. Has received prior therapy with TAS-102.
3. Is contraindicated for pembrolizumab and/or TAS-102, or have severe hypersensitivity to any of those drugs and/or their excipients.
4. Has any unresolved ≥Grade 2 toxicity (per CTCAE v5.0) attributed to any prior therapies at the time of enrollment.
5. Has had major surgery within 2 weeks prior to first dose of study interventions.
6. Has known active central nervous system (CNS) metastases.
7. Has received radiotherapy for gastric cancer treatment within 2 weeks prior to the first dose of study drugs.
8. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Has participated has used an investigational device within 4 weeks prior to the first dose of study intervention.
11. Has a history of uncontrollable or significant cardiovascular disease.
12. Has active (significant or uncontrolled) gastrointestinal bleeding.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years.
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active, unresolved infection requiring systemic therapy.
16. Has a known history of Human Immunodeficiency Virus (HIV) infection.
17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Has had an allogenic tissue/solid organ transplant.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ib (DLT) | within first 6weeks
  Phase Ib (Lead-in safety cohort): Dose-limiting toxicity (DLT)
Phase Ib (RP2D) | within first 6weeks
  Phase Ib (Lead-in safety cohort): Recommended Phase 2 dose (RP2D)
Objective response rate (ORR) | 6months after the last treatment of the last subject
  The proportion of patients in complete remission (CR) or partial remission (PR) among the best response (BOR) assessed by the investigator according to RECIST 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | 6months after the last treatment of the last subject
  Defined as the time start of study treatment until death by cause. Any subject not known to have died at the time of the analysis will be censored on the last recorded date on which the subject was known to be alive.
Progression-free survival (PFS) as assessed per RECIST 1.1 | 6months after the last treatment of the last subject
  Defined as the time from start of study treatment until the date of objective disease progression or death. Progression is defined in accordance with RECIST v1.1 criteria.
Disease control rate (DCR) as assessed per RECIST 1.1 | 6months after the last treatment of the last subject
  Defined as the proportion of subjects with a best objective response (BOR) of complete response (CR) or Partial response (PR), or stable disease maintained for a minium of twelve weeks from start of treatment, as defined by the RECIST 1.1.
Duration of response (DOR) as assessed per RECIST 1.1 | 6months after the last treatment of the last subject
  Defined as the time from the investigator's first determination of objective response to the first of disease progression or death according to RECIST 1.1.
Number of participants with Adverse Events that are related to treatment | Throughout the overall trial period as well as up to 3months after the last dose study treatment for each subject
  Safety and tolerability of the pembrolizumab and TAS-120 combination therapy as determined by adverse events categorized in accordance with CTCAE 5.0 Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG Rha, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No